CLINICAL TRIAL: NCT04886245
Title: Eye-Tracking FP "A Pilot Study of the Quantitative Evaluation of the Attention Paid to Faces With Facial Palsy by the Eye-tracking Technology.
Acronym: EyeTrackingFP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2019_843_0089
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Eye-tracking; Facial Palsy
Keywords: facial mimics; eye-tracking; Facial Palsy
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- facial palsy (Experimental): Patient with peripheral facial palsy, irrespective of grade, whether or not previously treated
  Interventions: Other: Video sequences
- healthy volunteers (Sham Comparator): - Subject without major facial sequelae
  Interventions: Other: Video sequences

INTERVENTIONS:
Other: Video sequences — videos will be made of each participant, during the realization of 5 movements that are the simple closure of the eyelids, the forced closure of the eyelids, the labial protrusion on the sound [o], the labial protrusion on the sound [pu] and the wide smile uncovering the teeth.
  Then, a video sequence will be realized thanks to the dedicated software Tobii Pro Lab®.

SUMMARY:
The facial palsy concerns between 15 and 40 people per 100000 inhabitants. They are of various etiologies such as infectious, tumoral, traumatic or idiopathic.

It has variable severities with sometimes heavy functional repercussions and different recovery potentials. The proposed palliative treatments are based on surgery, physiotherapy and botulinum toxin injections. However, when recovery is incomplete, acceptance is more difficult, with an impacted quality of life. In this context, patients' expectations and feelings about their care may become difficult for clinicians to apprehend.

The eye-tracking is widely used in the marketing field, but it also finds medical applications including head and neck lesions and facial palsy in particular. Published studies focus on the gaze of photographs, excluding any notion of dynamics and by the analysis of the gaze of outside observers, ignoring the patient's gaze.The main objective is to evaluate the attention paid to the facial side with abnormal facial movement by patients with facial paralysis compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* for patient with facial paralysis:
* Patient with peripheral facial palsy, irrespective of grade, whether or not previously treated
* Patient providing written informed consent
* Patient aged ≥ 18 years
* Patient affiliated to a social security system
* for Healthy voluntary subject :
* Subject without major facial sequelae
* Subject who provided written informed consent
* Major subject ≥ 18 years old
* Subject affiliated to a social security system

Exclusion Criteria:

* for Patient with facial paralysis:
* Patient with recent peripheral facial palsy whose total recovery is possible
* Patient unable to provide written informed consent
* Patient with difficulties to follow instructions and especially to stand in front of a computer screen
* Minor patient <18 years
* Patient under guardianship or curators or judicial safeguard
* for Healthy voluntary subject :
* Subject with major facial sequelae
* Subject not able to provide written informed consent
* Subject presenting difficulties in following instructions and in particular in standing still in front of a computer screen
* Minor subject < 18 years old
* Subject under guardianship or curators or judicial safeguard

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Variation of facial fixation day number between facial palsy patients and healthy volunteers | 30 days
Incidence of facial movement abnormality between facial palsy patients and healthy volunteers | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No